CLINICAL TRIAL: NCT05040763
Title: A Multi-Center Evaluation of Buccal Swabs With the Abbott ID NOW COVID-19 for Point-of-Care Detection SARS-CoV-2 in Pediatric Emergency Departments
Brief Title: PERC Health Canada COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REB21-1373
Record Dates: First submitted 2021-09-08; First posted 2021-09-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The primary objective of this study is to determine whether buccal swabs analyzed with the Abbott ID Now perform acceptably compared to standard of care COVID-19 swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 Swab Collection (Experimental): All participants will receive standard of care COVID-19 testing in addition to buccal swab COVID-19 testing
  Interventions: Diagnostic Test: Buccal Swabc- Copan flocked swab; Diagnostic Test: Standard of Care COVID-19 swab

INTERVENTIONS:
Diagnostic Test: Buccal Swabc- Copan flocked swab — All participants will have a buccal swab sampled collected from the inside of the mouth either by themselves or by their caregiver
Diagnostic Test: Standard of Care COVID-19 swab — All participants will receive a standard of care COVID-19 swab collected by a qualified healthcare professional

SUMMARY:
Although there are several licensed vaccines for SAR-CoV-2 (COVID-19) in Canada, none of them are approved for use in children under the age of 12, leaving five million children under 12 years unvaccinated. There is a need to find methods of mass rapid point of care testing in unvaccinated populations such as in schools that can be performed by a lay individual. This multi-center study will evaluate the clinical sensitivity of buccal swabs with the ID NOW COVID-19 device in comparison to standard of care COVID-19 testing at 15 pediatric emergency centres across Canada.

DETAILED DESCRIPTION:
This study will enroll approx 2882 participants under the age of 18 at 15 pediatric emergency centres across Canada. The purpose of the study is to evaluate the clinical sensitivity of buccal swab testing using Abbott ID NOW COVID-19device to detect SARS-CoV-2 infection among children aged 0-<18.0 years old presenting to the emergency department with an indication for SARS-CoV-2 testing as determined by the clinical care team. The study also seeks to identify factors that influence the accuracy of the testing approach and to examine the feasibility and perception of self/caregiver buccal swab sample collection.

In this prospective study, we will validate a self collected buccal swab that is analyzed with the Abbott ID NOW COVID-19 device against a reference RT-PCR nasal, nasopharyngeal (NP) or throat swab (or others) deemed standard of care at participating sites. The standard of care swabs will be collected by a qualified health professional and assessed by local laboratory services.

Individuals presenting to the emergency department that are identified as meeting the criteria as per local guidelines to be tested for SARS-CoV-2 (i.e. droplet precautions) will be appropriately consented and screened for participation in the study.

Eligible, consented participants will have their past medical history, COVID-19 symptom assessment, vaccination status, and physical exam findings collected from their charts.

A qualified healthcare professional will obtain a standard of care RT-PCR Swab from the participant. The results from this swab will be collected from the participants chart once available.

Depending on age, the study team will then train the participant/caregiver how to perform and obtain a buccal swab from the inside of the cheek. The collected buccal swab will be analyzed by the study team using the Abbott ID NOW COVID-19 device and results obtained within approx 15 mins.

Participants and their families will be notified of the qualitative result from the buccal swab.

Participants and their caregivers will be asked to complete pain assessment and acceptability questionnaires for both the standard of care and buccal swab tests.

ELIGIBILITY:
Inclusion Criteria:

1. Age <18.0 years old
2. Presenting to a participating emergency department
3. Consented to undergo local standard of care SARS-CoV-2 test
4. Able to read/speak English or French

Exclusion Criteria:

1. Inability or unwillingness of individual or legal guardian/representative to give written informed consent or child to give assent.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7263 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Buccal Swab Clinical Sensitivity | 3 month recruitment timeframe
  The study will evaluate the clinical sensitivity of buccal swab testing using Abbott ID NOW COVID-19 to detect SARS-CoV-2 infection among children aged 0-<18.0 years old presenting to the emergency department with an indication for SARS-CoV-2 testing as compared to standard of care reference standard COVID-19 swab testing

SECONDARY OUTCOMES:
Accuracy of Testing Approach | 3 month recruitment timeframe
  The team will Identify factors which influence the accuracy of testing such as symptoms onset, duration of symptoms, age, past medical history, vaccination status etc.
Feasibility and Acceptability of Buccal Swab Collection | 3 month recruitment timeframe
  The study will examine the feasibility and perception of self/caregiver buccal swab sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — University of Calgary
Locations (13):
- Canada (13):
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Hamilton, Ontario
  - McMaster Children's Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Laval, Québec, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Freedman SB, Kim K, Freire G, Kanngiesser A, Kam A, Doan Q, Wright B, Bhatt M, Berthelot S, Gravel J, Burstein B, Emsley J, Mater A, Porter R, Poonai N, Reddy D, Webster RJ, Goldfarb DM, Leifso K, Zemek R; Pediatric Emergency Research Canada (PERC) COVID Study Group. Accuracy of point-of-care SARS-CoV-2 detection using buccal swabs in pediatric emergency departments. Microbiol Spectr. 2024 Oct 29;12(12):e0188424. doi: 10.1128/spectrum.01884-24. Online ahead of print. PMID 39470284